CLINICAL TRIAL: NCT02628964
Title: Assessing the Use of Electronic Cigarettes (E-cigarettes) as a Harm Reduction Strategy
Brief Title: Electronic Cigarettes (E-cigarettes) as a Harm Reduction Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14-01178
Record Dates: First submitted 2015-09-28; First posted 2015-12-11 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Tobacco Use Disorder; Smoking
Keywords: smoking; cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 4.5% e-cig (Active Comparator): e-cigarettes with nicotine cartridges
  Interventions: Device: e-cigarettes
- 0 mg e-cig (Placebo Comparator): e-cigarettes with placebo cartridges (0mg).
  Interventions: Device: e-cigarettes

INTERVENTIONS:
Device: e-cigarettes — Participants and research assistants will be blind to the allocation of nicotine or placebo e-cigarettes as there are no difference in appearance or odor of the mist emitted from the e-cigarettes with and without nicotine containing cartridges.

SUMMARY:
The purpose of this study is to examine the feasibility of using e-cigarettes as a method for harm reduction and the effects of providing e-cigarettes (or placebo e-cigarettes) on smoking outcomes. Participants will be randomized to receive either e-cigarettes with nicotine cartridges or e-cigarettes with placebo cartridges, and followed for 3 weeks.

DETAILED DESCRIPTION:
This pilot study will be a two-arm, randomized controlled trial. The investigator will randomize 40 participants into each intervention arm. Participants will be randomized to one of the two arms: e-cigarettes with nicotine cartridges or e-cigarettes with placebo cartridges (0mg). Participants and research assistants will be blind to the allocation of nicotine or placebo e-cigarettes as there are no difference in appearance or odor of the mist emitted from the e-cigarettes with and without nicotine containing cartridges. Participants will be asked to track their nicotine use via text message. All participants will receive a 20-30 minute behavioral counseling consultation with a trained tobacco counselor. Counselors will review each participant's smoking pattern and offer tailored behavioral and environmental change strategies including specific smoking reduction strategy options. Participants will be given a supply of e-cigarettes and followed for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* 21-35 years old
* daily smokers who smoke at least 10 cigarettes per day (CPD)
* interested in reducing CPDs
* able to provide consent
* Use a cell phone and are willing/able to receive and respond to daily text messages regarding their cigarette use and e-cigarette use on their cell phone
* Willing to use an e-cigarette for 3 weeks

Exclusion Criteria:

* pregnant and/or breast feeding
* currently using smoking cessation medications (including other forms of Nicotine Replacement Therapy (NRT), buproprion, or varenicline)
* enrolled in a smoking cessation program or another cessation trial
* have used an e-cigarette in the past 14 days
* have used any other tobacco products (pipe, cigar, cigarillos, snuff, chewing tobacco, rolling tobacco, or hookah/shisha) in the past 30 days
* score ≥7 (men) or ≥5 (women) on the Alcohol Use Disorders Identification Test (AUDIT-C),
* score ≥ 5 on the Drug Abuse Screening Test-10 (DAST)
* report having a history of asthma, other airways diseases, or heart disease.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4.5% E-cig | 0 mg E-cig
Started | 50 | 50
Completed | 50 | 49
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4.5% E-cig | 0 mg E-cig | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 49 | 99
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 34 | 33 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic African American/black | 16 | 14 | 30
  Non-Hispanic white | 17 | 12 | 29
  Other non-Hispanic | 5 | 9 | 14
  Hispanic of any race | 11 | 13 | 24
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Number of Cigarettes Per Day (CPD)
Time Frame: Baseline up to 3 weeks
Measure: Mean (Standard Deviation); unit: cigarettes per day (CPD)
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 50 | 49
cigarettes per day (CPD) | 8.2 (5.1) | 7.3 (4.9)

2. Primary Outcome: Proportion of Participants Who Achieve 50% Reduction in Number of Cigarettes Per Day at 3 Weeks.
Description: Using the percent difference in number of cigarettes per day from baseline to 3-weeks, the proportion of participants who reduced their cigarette usage per day by 50% or greater
Time Frame: up to 3 weeks
Measure: Number; unit: proportion of participants
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 40 | 39
proportion of participants | .7 | .49

3. Secondary Outcome: Percent of Participants in Each Arm Who Reported Side Effects
Description: Percentage of participants who responded yes to a yes/no question about experiencing any side effects
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 40 | 39
percentage of participants | 22.5 | 10.5

4. Secondary Outcome: Number of Participants Using Additional Tobacco Products and/or Marijuana
Time Frame: Up to 12 weeks
Population: no data were collected for this Outcome Measure
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage Satisfaction Rating for the E-cigarettes
Description: Percent of participants who reported either "Strongly Agree" or "Agree" to liking using e-cigarettes at 3-weeks
Time Frame: 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 39 | 40
percentage of participants | 65 | 71.8

6. Secondary Outcome: Number of Nicotine Urges/Cravings
Time Frame: Up to 12 weeks
Population: no data were collected for this Outcome Measure
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing Withdrawal Symptoms
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: Up to 12 weeks
Population: no data were collected for this Outcome Measure
Arm/Group | 4.5% E-cig | 0 mg E-cig
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 Weeks
Arm/Group | 4.5% E-cig | 0 mg E-cig
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02628964/Prot_SAP_000.pdf